CLINICAL TRIAL: NCT05258786
Title: Pre-labor Ultrasound as a Visual Biofeedback Device for Maternal Pushing Education and Pelvic Floor Training - a Randomized Control Trial
Brief Title: Pre-labor Ultrasound as a Visual Biofeedback Device for Maternal Pushing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AU-HEA-NBA-20211128 Pre_labor
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy Related; Delivery Complication
Keywords: pre-labor education; biofeedback; ultrasound; vaginal delivery; fear of childbirth

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will collect the data from the files without knowing the participant's groups (intervention/control/standard care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): Transabdominal ultrasound will be applied to optimize the training program of contracting pelvic floor muscles, aiming to decrease postpartum urinary and fecal incontinence. Transperineal ultrasound will be used for pre-labor-coached maternal pushing aiming to improve pushing during the second stage of labor, reduce operative deliveries, the incidence of perineal tears, and urinary and fecal incontinence.
  Interventions: Behavioral: Pre-labor ultrasound as a visual biofeedback device for maternal pushing education and pelvic floor training
- Control group (No Intervention): A pelvic floor physiotherapist will provide the participants with a verbal explanation of how to contract pelvic floor muscles. without ultrasound.
- Standard care (No Intervention): Questionnaires only at four timeline points - before delivery at recruitment (T0), a week later (T2), immediately postpartum (T3), and two months postpartum (T4)

INTERVENTIONS:
Behavioral: Pre-labor ultrasound as a visual biofeedback device for maternal pushing education and pelvic floor training — 1. Ultrasound examination with the screen turned to the provider will assess the bladder movements at rest and during contraction of the pelvic floor and fetal head descent at rest and during pushing.
  2. The provider will turn the screen to the patient and explain the anatomical landmarks: bladder, fetal head, birth canal direction.
  3. A repeat of the first stage (1) with the screen turned to the patient: the biofeedback process. Bladder displacement will serve as a marker of pelvic floor contraction, and the delta in the progression angle will serve as a marker for effective pushing.
  4. Finally, the provider will turn the screen again from the patient and repeat the first stage.
  Arms: Intervention group

SUMMARY:
The study will observe the effect of antenatal biofeedback with transperineal and abdominal ultrasound applied by a pelvic floor physical therapist. The training will focus on pelvic floor training and maternal-coached pushing with ultrasound-based visual biofeedback. The investigators aim to assess maternal and neonatal obstetrical outcomes, urinary and fecal incontinence, and maternal psychological effects.

DETAILED DESCRIPTION:
Childbirth is a challenging process both emotionally and physically. The anxiety and anticipation accompanying pregnancy, labor, and delivery were reported to be relieved by pre-labor education, providing knowledge regarding the physiological process of labor to future parents.

Ultrasound examination enables the laboring women the opportunity to see fetal head movements in response to maternal pushing, and previous studies have revealed the physiological and psychological advantages of ultrasound-mediated intrapartum biofeedback during the second stage of labor.

Pre-labor sonographic maternal coaching has the advantage of a clean setting, avoiding the stressful, frequently hectic nature of labor and delivery wards, and may enable a more comprehensive implementation of the method, a structured training program, and better physical and psychological outcomes. All available literature regarding the application of intrapartum and pre-labor ultrasound refers to the examination performed by obstetricians.

The study will observe the effect of antenatal biofeedback with transperineal and abdominal ultrasound applied by a pelvic floor physical therapist. The training will focus on two aspects: pelvic floor training and maternal coached pushing - both with ultrasound-based visual biofeedback. The investigators aim to assess maternal and neonatal obstetrical outcomes, urinary and fecal incontinence, and maternal psychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* pregnant nullipara women with a low-risk pregnancy who are planned for vaginal delivery. The biofeedback will occur at 36-42 gestational weeks.

Exclusion Criteria:

* an inability to fill questionaries due to communication issues or cesarean section performed due to major obstetrical events.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2024-01-28 (Actual); Study Completion 2024-01-28 (Actual)

PRIMARY OUTCOMES:
length of the second stage of labor | up to 1 week after labor
  measure by time (min/hour)

SECONDARY OUTCOMES:
Mode of delivery | up to 1 week after labor
  Number of Participants with spontaneous vaginal or operative delivery (operative assisted - vacuum-assisted, forceps assisted, cesarean delivery)
Perineal tears | up to 1 week after labor
  Number of Participants with Perineal tears, specifically OASIS - obstetric anal sphincter Number of Participants with injuries
Urinary and fecal incontinence | up to 1 week after labor, and 2 month after labor.
  Number of Participants with Urinary and/ or fecal incontinence
Fear of birth questionnaire | Baseline, a week later , 1 week after labor and two months after labor
  6-36, higher score mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Noa Ben Ami, PhD, Principal Investigator — Ariel University
Locations (1):
- Noa Ben Ami, Ariel, Israel

IPD SHARING:
Plan to Share IPD: No